CLINICAL TRIAL: NCT07313891
Title: A Phase 3, Randomized Study Evaluating the Efficacy and Safety of NDV-01 Versus Observation in Participants With Intermediate-risk Non-muscle Invasive Bladder Cancer (BOOST)
Brief Title: A Study of Adjuvant NDV-01 (Sustained-release Gemcitabine-docetaxel) for the Treatment of Intermediate Risk NMIBC Following TURBT
Acronym: BOOST
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REL-NDV01-301
Record Dates: First submitted 2025-12-29; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer Superficial (Non-Invasive); Bladder (Urothelial, Transitional Cell) Cancer; Urothelial Carcinoma Bladder; Urologic Cancer
Keywords: NMIBC; non-muscle-invasive bladder cancer; bladder cancer
MeSH Terms: conditions — Neoplasms; Urologic Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: A Phase 3, Open-label Randomized Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: NDV-01 (sustained-release gemcitabine-docetaxel) (Experimental): Intervention with NDV-01 (sustained-release gemcitabine-docetaxel)
  Interventions: Drug: NDV-01 (sustained-release gemcitabine-docetaxel)
- Arm B: surveillance (No Intervention): Surveillance with Cystoscopy, Urine Cytology, Biopsy (if indicated)

INTERVENTIONS:
Drug: NDV-01 (sustained-release gemcitabine-docetaxel) — Intravesical instillation of NDV-01 (sustained-release gemcitabine-docetaxel)
  Arms: Arm A: NDV-01 (sustained-release gemcitabine-docetaxel)

SUMMARY:
This is a Phase 3, open-label, randomized trial designed to evaluate the DFS of TURBT followed by NDV-1 (sustained-release gemcitabine-docetaxel) versus TURBT followed by surveillance for the treatment of participants with IR-NMIBC.

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to NDV-1 (sustained-release gemcitabine-docetaxel) after TURBT (Arm A) vs surveillance after TURBT (Arm B).

Participants in Arm A will receive an induction course and then monthly maintenance courses of NDV-1 (sustained-release gemcitabine-docetaxel) through Month 12, if there is no disease recurrence.

Disease status will be assessed using urine cytology, cystoscopy, and directed TURBT/biopsy (if indicated) every 3 months for the first 2 years after randomization and then every 6 months for an additional year or until disease recurrence.

Participants in Arm B who recur with IR-NMIBC after TURBT and surveillance will be offered treatment with NDV-1 (sustained-release gemcitabine-docetaxel) as per the treatment schedule in Arm A.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed diagnosis (within 90 days of randomization) of IR NMIBC based on the AUA/SUO criteria of IR NMIBC.
2. Participants must have ≥ 1 IBCG risk factors: multiple tumors, early recurrence (Within 1 year), frequent recurrences (> 1 per year), tumor size (> 3 cm), failure of prior intravesical therapy.
3. Visible papillary disease must be fully resected prior to randomization, and absence of disease must be documented at Screening cystoscopy. The same method for visualizing disease at Screening cystoscopy should be used throughout for the participant (white light versus enhanced assessment method).
4. Patients with LG T1 may be eligible after repeat-TURBT (within 4 weeks of first TURBT) if the repeat pathology shows non-invasive (Ta or less) or no disease. Original and repeat-TURBT must confirm that muscularis propria is present and uninvolved in the specimen. TURBT to occur within 4 months of screening. All pathology specimens must be predominantly urothelial (transitional cell) and have less than 20% variant (e.g., sarcomatoid, squamous component) histology.

Exclusion Criteria:

1. Histologically confirmed diagnosis of HR NMIBC (including CIS) or MIBC, locally advanced, nonresectable, or metastatic urothelial carcinoma at any time prior to enrollment.
2. Has had urothelial carcinoma outside of the urinary bladder, (including prostatic urethra, ureter, or renal pelvis) or has a predominant histological variant of UC. Ta/any T1, CIS of the upper urinary tract is allowable if treated with complete nephroureterectomy more than 24 months prior to initiating study.
3. Participant has tumor(s) involving the prostatic urethra (ductal or stromal).
4. N+ and/or M+ per CT/MR urography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
To compare DFS between study arms | From date of randomization to at least 2 years of follow-up assessing for DFS events.
  Time from randomization to either time of the first recurrence or progression, or death due to any cause, whichever occurs first. It is hypothesized that sustained local delivery of GEM and DOCE (via NDV-01) in participants with IR-NMIBC will result in longer DFS than achieved with observation after TURBT. Under the exponential distribution assumption for DFS, this translates into testing the statistical hypothesis that the hazard ratio is significantly less than 1.0. Primary endpoint will be tested using a one-sided 2.5% level of significance.
  This study will randomize 302 participants in a 1:1 randomization ratio. The primary efficacy analysis for DFS will be performed when approximately 133 DFS events have been observed. Assuming a 25% recurrence rate (hazard rate 0.14384) in the 2-year DFS in the treated arm, vs. a 40% recurrence rate (hazard rate 0.2554) in the control arm (i.e., a hazard ratio of 0.563 under the exponential distribution assumption for DFS, 53 vs. 80 events.

CONTACTS AND LOCATIONS:
Overall Officials: Raj S Pruthi, MD MHA, Study Director — Relmada Therapeutics

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant privacy concerns, limitations of informed consent, and regulatory and data governance constraints. De-identified aggregate results will be made publicly available through ClinicalTrials.gov and scientific publications.

REFERENCES:
- [Result] Tan WS, McElree IM, Davaro F, Steinberg RL, Bree K, Navai N, Dinney CP, O'Donnell MA, Li R, Kamat AM, Packiam VT. Sequential Intravesical Gemcitabine and Docetaxel is an Alternative to Bacillus Calmette-Guerin for the Treatment of Intermediate-risk Non-muscle-invasive Bladder Cancer. Eur Urol Oncol. 2023 Oct;6(5):531-534. doi: 10.1016/j.euo.2023.06.011. Epub 2023 Jul 18. PMID 37468392
- [Result] Holzbeierlein JM, Bixler BR, Buckley DI, Chang SS, Holmes R, James AC, Kirkby E, McKiernan JM, Schuckman AK. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline: 2024 Amendment. J Urol. 2024 Apr;211(4):533-538. doi: 10.1097/JU.0000000000003846. Epub 2024 Jan 24. PMID 38265030
- See also: AUA/SUO Guidelines for NMIBC — https://www.auanet.org/guidelines-and-quality/guidelines/bladder-cancer-non-muscle-invasive-guideline